CLINICAL TRIAL: NCT02545556
Title: HepaSphere Interventional Therapy Using Digital Subtraction Angiography（DSA）Combined With Cryosurgery for Liver Cancer: Clinical Trial
Brief Title: Liver Cancer HepaSphere Combined With Cryosurgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Liver hepaSphere cryosurgery
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2015-10

CONDITIONS: Liver Cancer
Keywords: Liver Cancer; HepaSphere; cryosurgery
MeSH Terms: conditions — Liver Neoplasms | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HepaSphere combined with cryosurgery (Experimental): liver cancer patients received HepaSphere interventional therapy using the digital subtraction angiography（DSA）combined with cryosurgery
  Interventions: Procedure: HepaSphere combined with cryosurgery
- control (Placebo Comparator): liver cancer patients received traditional therapy
  Interventions: Procedure: HepaSphere combined with cryosurgery

INTERVENTIONS:
Procedure: HepaSphere combined with cryosurgery — liver cancer patients received HepaSphere interventional therapy using the digital subtraction angiography（DSA）combined with cryosurgery

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of HepaSphere interventional therapy using digital subtraction angiography（DSA）combined with cryosurgery for liver cancer.

DETAILED DESCRIPTION:
By enrolling patients with liver cancer adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of HepaSphere interventional therapy using digital subtraction angiography（DSA） combined with cryosurgery for liver cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-80
2. Karnofsky performance status >60
3. Diagnosis of pancreatic cancer based on histology or the current accepted radiological measures.
4. Classification tumor,nodes,metastasis-classification(TNM) stage: Ⅱ,Ⅲ,Ⅳ
5. Will receive interventional therapy
6. Life expectancy: Greater than 3 months
7. Patients' routine blood test, liver function and kidney function have no obvious abnormalities
8. Ability to understand the study protocol and a willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients with other primary tumor except liver cancer
2. History of coagulation disorders or anemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse events | 1 year

SECONDARY OUTCOMES:
Percentage of lesions interventional therapy that show no sign of recurrence 12 months after | 1 year
Progress free disease (PFS) | 1 year
Overall survival (OS) | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Niu, PhD, Study Chair — Fuda Cancer Hospital
Locations (1):
- Central laboratory in Fuda cancer hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Niu L, Chen J, Yao F, Zhou L, Zhang C, Wen W, Bi X, Hu Y, Piao X, Jiang F, Zeng J, Liu W, Li J, He L, Mu F, Zuo J, Xu K. Percutaneous cryoablation for stage IV lung cancer: a retrospective analysis. Cryobiology. 2013 Oct;67(2):151-5. doi: 10.1016/j.cryobiol.2013.06.005. Epub 2013 Jun 24. PMID 23806858
- See also: related information — http://www.ncbi.nlm.nih.gov/pubmed/25937772